CLINICAL TRIAL: NCT05724875
Title: Randomized Phase II Selection Trial of FLASH Versus Conventional Radiotherapy for Patients with Localized Cutaneous Squamous Cell Carcinoma or Basal Cell Carcinoma
Brief Title: FLASH Radiotherapy for Skin Cancer
Acronym: LANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Prof. Olivier Gaide, MD-PhD, Prof, MD, PhD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-0024-LANCE-2020
Record Dates: First submitted 2023-01-17; First posted 2023-02-13 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Basal Cell Carcinoma; Cutaneous Squamous Cell Carcinoma
Keywords: FLASH therapy; basal cell carcinoma; cutaneous squamous cell carcinoma; high dose rate radiotherapy
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: FLASH RT (Experimental)
  Interventions: Device: FLASH RT
- Arm B: Conventional RT (Active Comparator)
  Interventions: Device: Conventional RT

INTERVENTIONS:
Device: FLASH RT — For T1 (small) lesions: 22 Gy single dose FLASH RT; For T2 (large) lesions: 5 x 6 Gy fractionated dose FLASH RT
  Other Names: High dose rate radiotherapy
  Arms: Arm A: FLASH RT
Device: Conventional RT — For T1 (small) lesions: 22 Gy single dose conventional RT; For T2 (large) lesions: 5 x 6 Gy fractionated dose conventional RT
  Arms: Arm B: Conventional RT

SUMMARY:
This is a single center randomized selected Phase II study of FLASH radiotherapy (RT) versus standard of care (SOC) radiotherapy in patients with localized Cutaneous Squamous Cell Carcinoma (cSCC) or Basal Cell Carcinoma (BCC).

In summary, the aims of the study are to describe and compare the toxicity and efficacy of high dose rate radiotherapy (FLASH therapy) to SOC conventional radiotherapy (according to the standard guidelines per lesion size) through a randomized Phase II selection study in patients presenting localized cSCC or BCC requiring a radiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed study Informed Consent Form
* Karnofsky Performance Status (KPS) ≥ 60
* Age ≥ 60 years
* Patients with histologically proven cSCC or patients with BCC either histologically proven or proven by non-invasive imaging: either Optical Coherence Tomography (OCT), Line-field OCT (LC-OCT) or Reflectance Confocal Microscopy (RCM)
* Patients requiring radiotherapy treatment according to the dermato-oncology tumor board: patients who cannot undergo surgical procedure or patients who decline surgical resection, and/or anatomical locations where surgery can compromise function or cosmesis.
* T1-T2 N0 lesions with a small (T1; lesion ≤ 2cm in diameter) or large (T2; 2cm < lesion ≤ 4 cm) volume (TNM Classification of Malignant Tumours (TNM) Union for International Cancer Control (UICC), 8th Edition)
* Lesions should be at least 4 cm apart if treated with 2 different modalities (including surgical treatment of lesions). Lesions should not be located on the face, except on the forehead, above a line situated 1 cm above the eyebrows. Lesions located on the scalp can be treated.

Exclusion Criteria:

* Previous radiotherapy in the treated area
* Concomitant auto-immune disease with skin lesions
* Concomitant use of radio-sensitizer drug
* Cognitive disorders not compatible with the signature of informed consent or that may compromise compliance with the requirements of the study
* Current, recent (within 10 days prior to start of study treatment), or planned participation in an experimental drug study (before end of treatment (EOT) visit)
* Concomitant use of systemic chemotherapy for a cancer other than the skin cancer(s)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of ≥ grade 3 skin toxicity adverse events (AEs) according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | up to 6 weeks after radiotherapy
  To evaluate the safety of FLASH radiotherapy measured by the collection of ≥ grade 3 skin toxicity AEs according to CTCAE version 5.0. The severity of a specific event is graded i.e. mild (grade 1), moderate (grade 2), severe (grade 3), life-threatening (grade 4), or death (grade 5) using the CTCAE Grading Table.
Hierarchically tested efficacy measured by local control rate | From Day 1 up to 12 months post-treatment
  At day 1, 21, 28, 42, and months 3, 6, and 12 post-treatment, the investigator will measure (with a caliper) the largest diameter of selected lesions for irradiation.
  Tumor response of each irradiated lesion will be assessed by the investigator as follow:
  * Complete Response: the irradiated lesion is no more visualized
  * Partial Response: the irradiated largest lesion dimension decreased by 30% at least from baseline (day 1)
  * Progressive Disease: the irradiated largest lesion dimension increased by 20% at least from baseline (day 1)
  * Stable Disease: no Complete Response, no Partial Response, no Progressive Disease

SECONDARY OUTCOMES:
Frequency of acute side effects observed "in radiation field" | up to 3 months after radiotherapy
Frequency of late side effects observed "in radiation field" | from ≥ 3 months after radiotherapy until 12 months post-treatment start
Evaluation of tumor response | From Day 1 up to 12 months post-treatment
  Blinded Imaging Central Review (BICR) of photographs will evaluate tumor response by grading the size of the residual tumor in comparison to the size of the tumor on the day of irradiation (in percentage). 0% means no residual tumor and treatment success, 100% or more indicate a total lack of tumor response.
  A baseline photograph will be taken the day of the treatment (day 1) in a pre-therapeutic setting with skin delineation of the lesion. Then photos will be repeated at day 21 (+/-2d), day 28 (+/-2d), day 42 (+/-3d) after treatment, then at 3 (+/-7d), 6 (+/-14d), 12 (+/-14d) months after treatment, and at progression.
Evaluation of "in radiation field" normal tissues reaction around the treated tumors | From Day 1 up to 12 months post-treatment
  Blinded Imaging Central Review (BICR) of photographs will evaluate "in radiation field" normal tissues reaction around the treated tumors by grading radiation induced skin reactions, grade 1-5, using the CTCAE scale.
  A baseline photograph will be taken the day of the treatment (day 1) in a pre-therapeutic setting with skin delineation of the lesion. Then photos will be repeated at day 21 (+/-2d), day 28 (+/-2d), day 42 (+/-3d) after treatment, then at 3 (+/-7d), 6 (+/-14d), 12 (+/-14d) months after treatment, and at progression.
Epidermis thickness measured by Optical coherence tomography (OCT) | at baseline, at 4 weeks, at 6 months, and at 12 months post-treatment
  Epidermis thickness in micrometer will be measured by OCT and compared between irradiated skin and normal non-irradiated skin
Epidermis roughness measured by OCT | at baseline, at 4 weeks, at 6 months, and at 12 months post-treatment
  Epidermis roughness in micrometer will be measured by OCT and compared between irradiated skin and normal non-irradiated skin
Plexus depth measured by OCT | at baseline, at 4 weeks, at 6 months, and at 12 months post-treatment
  Plexus depth in micrometer will be measured by OCT and compared between irradiated skin and normal non-irradiated skin
Vessel density measured by OCT | at baseline, at 4 weeks, at 6 months, and at 12 months post-treatment
  Vessel density, expressed as percent of the surface covered by the vessels in the examined area, will be measured by OCT and compared between irradiated skin and normal non-irradiated skin
Size of vessels measured by OCT | at baseline, at 4 weeks, at 6 months, and at 12 months post-treatment
  Mean size (in micrometer) of all vessels in the examined area will be measured by OCT and compared between irradiated skin and normal non-irradiated skin
Number of hairs counted by OCT | at baseline, at 4 weeks, at 6 months, and at 12 months post-treatment
  Number of hairs in the examined area will be counted by OCT and compared between irradiated skin and normal non-irradiated skin
Size of hairs measured by OCT | at baseline, at 4 weeks, at 6 months, and at 12 months post-treatment
  Mean size (in micrometer) of all hairs in the examined area will be measured by OCT and compared between irradiated skin and normal non-irradiated skin

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Gaide, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois; Jean Bourhis, MD, PhD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland